CLINICAL TRIAL: NCT04305834
Title: A Phase IIA Trial Assessing the Tolerability of Abemaciclib in Combination With Endocrine Therapy in Patients Age 70 and Older With Hormone Receptor Positive Metastatic Breast Cancer Who Have Progressed on or After Prior CDK 4/6 Inhibition
Brief Title: Abemaciclib and Endocrine Therapy in Older Patients With Breast Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19206; NCI-2019-08847 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19206 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-03-02; First posted 2020-03-12 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Hormone Receptor Positive Breast Carcinoma; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (abemaciclib) (Experimental): Patients receive abemaciclib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY-2835219; LY2835219; Verzenio
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase IIa trial studies the side effects of abemaciclib monotherapy in treating patients age 70 years and older with hormone receptor positive, HER2 negative breast cancer that has spread to other places in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the incidence of grade 3 or higher toxicities attributed to abemaciclib monotherapy in adults aged 70 or older with hormone receptor positive metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To describe the full toxicity profile including all grade 2 and higher adverse events, and patient-reported adverse events (AEs) using Patients Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE) measures.

II. To describe rates of dose reductions, dose holds, treatment discontinuations due to factors other than progression, and hospitalizations.

III. To estimate median (and 95% confidence interval [CI]) failure-free survival, progression-free survival and overall survival.

IV. To describe the results of Was It Worth It (WIWI) and Overall Treatment Utility (OTU) questionnaires.

V. To describe the rate of adherence to abemaciclib. VI. To determine average plasma steady-state abemaciclib Ctrough concentrations.

VII. To evaluate the association of adherence rate with abemaciclib plasma t-rough concentrations.

VIII. To describe associations between cancer-specific, comprehensive Geriatric Assessment (cGA) scores and the incidence of toxicities and their grade.

EXPLORATORY OBJECTIVE:

I. To determine the association between biomarkers of aging and grades 3 or higher toxicity.

OUTLINE:

Patients receive abemaciclib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* Age >= 70 years
* Life expectancy > 6 months
* Ability to read and understand English or Spanish
* Measurable or non-measurable disease
* Histologically or cytologically confirmed diagnosis of:

  * Estrogen-receptor positive and/or progesterone receptor positive breast cancer determined by immunohistochemistry (IHC) methods according to the local institution standard protocol
  * HER2-negative breast cancer defined as negative if the IHC status is 0 or 1+, or if IHC is 2+ and in situ hybridization assay is negative per American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines
* Radiographically confirmed metastatic breast cancer
* Progressed on prior endocrine therapy or palbociclib or ribociclib or chemotherapy
* Patients who received chemotherapy recovered from the acute side effects to prior cancer therapy (except alopecia or residual grade 2 peripheral neuropathy) to =< grade 1 or baseline. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy)
* Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization
* Absence of central nervous system (CNS) involvement unless they meet ONE of the following criteria:

  * Untreated brain metastases (e.g., lesions < 1 cm) not needing immediate local therapy
  * Previously treated brain metastases not needing immediate local therapy

    * At least 4 weeks from the last date of prior therapy completion (including radiation and/or surgery) to starting the study treatment
    * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases
* Absence of interstitial lung disease/pneumonitis
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 8 g/dL

  * (Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion)
* In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 x upper limit of normal (ULN)

  * If the patient has liver metastases, ALT and AST < 5 x ULN
* In patients without Gilbert's syndrome, total bilirubin =< 1.5 x ULN; In patients with Gilbert's syndrome, total bilirubin =< 2.0 x ULN or direct bilirubin within normal limits (WLN)
* Creatinine clearance of >= 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula

Exclusion Criteria:

* Major surgery within 14 days prior to receiving study drug or has not recovered from major side effect
* Patient is currently receiving any of the prohibited medications detailed below and cannot be discontinued 7 days prior to starting study drug

  * Other investigational therapy should be given to participants
  * Anticancer agents other than the study medications administered as part of this study protocol should be given to participants. If such agents are required for a participant then the participant must first be withdrawn from the study
  * Co-medication that may interfere with study results; e.g. immune-suppressive agents other than corticosteroids, such as systemic cyclosporine and tacrolimus are prohibited during the treatment phase of the study, unless discussed with principal investigator felt to be of low clinical risk to the participant
  * Use of herbal medications may have unknown interactions with the metabolism of the study agents, and therefore are prohibited from use during the treatment phase of the trial
* Known hypersensitivity to any of the excipients of abemaciclib
* Active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C (for example, hepatitis B surface antigen positive). Screening is not required for enrollment
* Impairment of gastrointestinal (GI) function or GI disease that in the investigator's opinion may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* History of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* Patient has any other concurrent severe or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis)
* Inability to swallow oral medications
* Serious or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance < 30 ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea)
* History of non-compliance to medical regimen
* Patients with a prior malignancy diagnosed within 2 years and with evidence of disease (except adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2026-08-21 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher toxicities | Up to 30 days post treatment
  Adverse events will be characterized using the descriptions and grading scales found in the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v). 5.0.

SECONDARY OUTCOMES:
Incidence of toxicities | Up to 30 days post treatment
  Toxicities will be graded and named according to CTCAE v. 5.0.
Incidence of toxicities | Up to cycle 6
  Toxicities will be captured by Patient Reported Outcome (PRO)-CTCAE.
Dose reductions | Up to cycle 6
  Will assess rates of dose reductions.
Dose holds | Up to 30 days post treatment
  Will assess rates of dose holds.
Treatment discontinuations due to factors other than progression | Up to 30 days post treatment
  Will assess rates of treatment discontinuations.
Hospitalizations | Up to 2 years post treatment
  Will assess rates of hospitalizations.
Time to end of treatment | Up to end of treatment
  Will estimate median (and 95% confidence interval [CI]) failure-free survival using Kaplan-Meier estimates and through Cox regression to adjust for covariates.
Progression free survival | Up to 2 years post treatment
  Will estimate median (and 95% CI) progression-free survival using Kaplan-Meier estimates and through Cox regression to adjust for covariates.
Overall survival | Up to 2 years post treatment
  Will estimate median (and 95% CI) overall survival using Kaplan-Meier estimates and through Cox regression to adjust for covariates.
Was It Worth It (WIWI) response | Up to end of treatment
  Will be assessed using the WIWI questionnaire.
Overall treatment utility (OTU) response | Up to end of treatment
  Will be assessed using the OTU questionnaire.
Adherence to abemaciclib | Up to end of treatment
  Adherence defined as taking 90% of scheduled doses per cycle. Scheduled doses are assigned doses for the participant which may vary per participant depending on whether or not there a hold in treatment. Adherence will be calculated based on consolidation of pill diary with returned unused pills, and, for City of Hope (COH) Duarte patients, Medication Event Monitoring bottle caps.
Average plasma steady-state abemaciclib C-trough concentrations | Up to 2 years post treatment
Pharmacokinetic (PK) parameter of plasma trough concentration | Up to 2 years post treatment
  Will evaluate the association of adherence rate with abemaciclib plasma trough concentrations.
Geriatric assessment scores | Up to 2 years post treatment
  Domains include: functional status, co-morbid medical conditions, cognitive function, nutritional status, social support and psychological state, and a review of medications.
Incidence of toxicities attributable to agent | Up to 2 years post treatment
  Graded by CTCAE v 5.0.

OTHER OUTCOMES:
Biological age via deoxyribonucleic acid (DNA) methylation level | Up to 2 years post treatment
Genome-wide methylome and transcriptome analyses | Up to 2 years post treatment
Incidence of toxicities at least possibly attributable to agent | Up to 2 years post treatment
  Graded by CTCAE v 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York